CLINICAL TRIAL: NCT06290180
Title: Healing Lodge First Face Training Evaluation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge Health Alliance (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Heather Gray, Director of Academic Affairs, Division on Addiction, Cambridge Health Alliance
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 13632; 1S06GM146095 (NIH)
Record Dates: First submitted 2024-02-13; First posted 2024-03-04 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Addiction; Depression/Anxiety; Trauma, Psychological; Self-harm
Keywords: mental health; prevention; addiction; substance use disorders
MeSH Terms: conditions — Behavior, Addictive; Depression; Anxiety Disorders; Psychological Trauma; Self-Injurious Behavior; Psychological Well-Being; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Pre/post/3-month follow-up model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healing Lodge First Face Training Evaluation Study (Experimental): All participants in this evaluation will be assigned to the First Face for Mental Health training condition. The investigators will use a pre-post design to measure change in relevant outcomes from pre-training, to post-training, to 3-months post-training.
  Interventions: Behavioral: First Face for Mental Heatlh

INTERVENTIONS:
Behavioral: First Face for Mental Heatlh — First Face for Mental Health is a culturally-appropriate community-based mental health training for lay persons and others that prepares learners to provide assistance to someone having a mental health crisis. The course takes approximately 8 hours to complete.

SUMMARY:
The purpose of this study is to evaluate a culturally grounded training program, xaʔtus (meaning First Face) for Mental Health. This program will train community members in how to recognize and respond to youth and adults experiencing mental health crises and ways to serve as a bridge between these individuals and the help they need. All Healing Lodge staff are being asked to complete First Face training.

To evaluate First Face, the investigators will ask all trainees to complete surveys before and after training, and again 3 months later. These surveys will measure knowledge about mental health and addiction, as well as the ability and confidence to respond appropriately to mental health crises. The study will help the investigators understand whether the First Face training program influences mental health and attitudes, as well as responses to mental health crisis situations.

DETAILED DESCRIPTION:
With funding from the National Institutes for Health, the investigators created First Face for Mental Health. First Face is a culturally-appropriate community-based mental health training that prepares trainees to provide assistance to someone having a mental health crisis. The more community members within Tribal nations who are trained in a culturally sensitive program to provide support to youth in recovery and members struggling with mental health problems or crises, the better positioned that community is to create a supportive recovery environment for its youth. The investigators are in the process of launching First Face trainings and evaluations among several Tribal communities. Additionally, they will be training staff from the Healing Lodge of the Seven Nations (HL) in the First Face program. This particular application concerns the evaluation of First Face training among HL staff. The investigators will measure primary and secondary outcomes at pre-training, post-training, and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Employment at the Healing Lodge of the Seven Nations
* Selection to participate in First Face for Mental Health training

Exclusion Criteria:

° Previous completion of First Face for Mental Health training

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Healing Lodge of the Seven Nations, Spokane Valley, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided
This study will be governed by a Data Sharing Agreement between the Healing Lodge of the Seven Nations and Cambridge Health Alliance. That Agreement is still pending.

REFERENCES:
- [Background] Watson AC, Miller FE, Lyons JS. Adolescent attitudes toward serious mental illness. J Nerv Ment Dis. 2005 Nov;193(11):769-72. doi: 10.1097/01.nmd.0000185885.04349.99. PMID 16260937
- [Background] Talbot JA, Ziller EC, Szlosek DA. Mental Health First Aid in Rural Communities: Appropriateness and Outcomes. J Rural Health. 2017 Jan;33(1):82-91. doi: 10.1111/jrh.12173. Epub 2016 Jan 28. PMID 26817852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Pre- and post-training data were collected in April and December, 2024. During 2024, the Healing Lodge employed 107 unique staff members. All were instructed that they were required to complete a First Face training. In total, 102 employees (95.3% of the year-round total) completed the First Face training. Not all trainees enrolled in the study. A total of 92 trainees in the study. Follow-up data were collected until April, 2025.
Pre-assignment Details: All participants were assigned to complete the First Face training; there was no comparison group.
Groups:
- Intervention group: All participants were assigned to receive the First Face for Mental Health training.
Period: Overall Study
Arm/Group | Intervention group
Started | 92
Completed | 47
Not Completed | 45

BASELINE CHARACTERISTICS:
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 92
Age, Customized [Count of Participants; unit: Participants] — We did not collect age data in this study. Population: As mentioned above, we did not collect age data in this study.
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Man | 41
  Gender: Woman | 47
  Gender: Another description | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Tribal membership: Enrolled in or descended from a federally-recognized Tribe | 32
  Tribal membership: Not enrolled in or descended from a federally-recognized Tribe | 60
Reside on a reservation [Count of Participants; unit: Participants]
  Reside on a reservation | 0
  Do not reside on a reservation | 92
Years working with at-risk youth [Mean (Standard Deviation); unit: Years] | 8.23 (8.98)
Department [Count of Participants; unit: Participants]
  Maintenance | 6
  Behavioral health | 44
  Administration | 13
  Medical | 5
  Mental health | 4
  Programs and support services | 16
  Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Attitudes Towards Serious Mental Illness - Adolescent Version
Description: The Attitudes Towards Serious Mental Illness - Adolescent Version (ATSMI-AV) is a validated 21-item self-report scale designed to measure attitudes towards mental illness. Participants respond on a 5-point Likert scale. The scale measures five aspects of mental health attitudes: threat, social construction/concern, wishful thinking, categorical thinking and out of control. The investigators will calculate an overall score as well as factor-specific scores, if they observe adequate internal reliability.
  Each item has response categories ranging from Completely disagree (coded as 1) to Completely agree (coded as 5), and a mean of all 21 items is calculated to create the scale. The scale has a possible range of 1 to 5 Higher scores indicate higher levels of stigma towards mental illness.
Time Frame: Included at pre-training, post-training (i.e. immediately after training), and 3-months post-training
Population: Some missing data, some participants lost to attrition.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 38
Score on a scale
  Pre-training | 2.05 (0.11)
  Post-training | 1.94 (0.10)
  3-month follow-up | 1.96 (0.11)

2. Primary Outcome: First Face Knowledge Assessment
Description: This is a 12-question quiz testing participants' knowledge of concepts taught in the First Face training. Some questions offer the opportunity to earn more than one point. The investigators will score each response as correct or incorrect and sum scores (possible range = 0-17) on each occasion. Higher scores indicate better knowledge of First Face concepts.
Time Frame: Included at pre-training, post-training (i.e. immediately after training), and 3-months post-training
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 39
Score on a scale
  Pre-training | 9.18 (0.42)
  Post-training | 13.04 (0.53)
  3-month follow-up | 12.26 (0.58)

3. Primary Outcome: Perceived Competence to Respond
Description: A 10-item measure that taps respondents' confidence in their competence to respond to and help people experiencing mental health problems (i.e., Confidence in Recognizing, Intervening and Connecting Individual(s) with Resources Scale). Each response option has a possible range of 1 (Not at all confident) to 5 (Very confident), and a mean score will be calculated from all 10 items to yield a scale with a possible range of 1 to 5. Higher values indicate greater perceived competence respond to and help people experiencing mental health problems.
Time Frame: Included at pre-training, post-training (i.e. immediately after training), and 3-months post-training
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 37
Score on a scale
  Pre-training | 4.17 (0.14)
  Post-training | 4.44 (0.09)
  3-month follow-up | 4.28 (0.13)

4. Secondary Outcome: Satisfaction With Training
Description: One item administered immediately post-training asking about satisfaction with training (from 1 ("very dissatisfied") to 7 ("very satisfied")), with higher scores indicating greater satisfaction.
Time Frame: Post-training (i.e. immediately after training)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 90
Score on a scale | 2.92 (1.98)

5. Secondary Outcome: Use of First Face Learnings
Description: Yes/no measure assessing whether participants used their training at all (in either personal or professional life) in the 3 months following training.
Time Frame: 3-months post-training
Population: Some missing data
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 46
Participants
  Missing | 1
  Yes-used training | 37
  No - did not use training | 9

6. Secondary Outcome: Intended Use of First Face Learnings in Personal Life
Description: Participants will report how likely they are to use the First Face training in the personal life on a 4-point scale from Not at all to To a great extent.
Time Frame: Post-training (i.e. immediately after training)
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 90
Participants
  Missing | 4
  Somewhat | 28
  To a great extent | 58
  Very little | 0
  Not at all | 0

7. Secondary Outcome: Intended Use of First Face Learnings in Professional Life
Description: Participants will report how likely they are to use the First Face training in the professional life on a 4-point scale from Not at all to To a great extent.
Time Frame: Post-training (i.e. immediately after training)
Measure: Count of Participants; unit: Participants
Arm/Group | Healing Lodge First Face Training Evaluation Study
Number analyzed (Participants) | 90
Participants
  Missing | 5
  Somewhat | 21
  To a great extent | 62
  Very little | 2
  Not at all | 0

ADVERSE EVENTS:
Time Frame: From enrollment until the end of follow-up, up to 3 months.
Description: No events to report.
Arm/Group | Healing Lodge First Face Training Evaluation Study
All-Cause Mortality (participants affected / at risk) | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90
Other Adverse Events (participants affected / at risk) | 0/90

LIMITATIONS AND CAVEATS:
Major limitations of this study include the lack of a comparison group and the lack of a longer-term follow-up. Future studies with more rigorous designs are needed before we can draw firm conclusions about the impact of First Face training, including whether positive effects on knowledge and perceived situational competence are sustained beyond the period immediately following training. Future research could compare First Face training against a waitlist control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/80/NCT06290180/Prot_002.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/80/NCT06290180/SAP_000.pdf
  • Informed Consent Form (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/80/NCT06290180/ICF_001.pdf